CLINICAL TRIAL: NCT01012492
Title: Safety and Tolerability Trial of Abatacept-based Immunosuppression for Prevention of Acute GvHD During Unrelated Donor Hematopoietic Stem Cell Transplant
Brief Title: Pilot of Abatacept-based Immunosuppression for Prevention of Acute GvHD During Unrelated Donor HCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Leslie Kean, MD, PhD, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00024488; Abatacept (Other: Other)
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Results first posted 2017-09-15 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-10

CONDITIONS: AML; ALL; Undifferentiated Leukemia; Biphenotypic Leukemia; Refractory Anemia; Refractory Anemia With Ringed Sideroblasts; Refractory Cytopenia With Multilineage Dysplasia; Ref. Cytopenia w Multilineage Dysplasia & Ringed Sideroblasts; Refractory Anemia With Excess Blasts-1 (5-10% Blasts); Refractory Anemia With Excess Blasts-2 (10-20% Blasts); Myelodysplastic Syndrome, Unclassified; MDS Associated With Isolated Del (5q)
Keywords: cancer; leukemia; transplant; bone marrow
MeSH Terms: conditions — Anemia, Refractory; Myelodysplastic Syndromes; Neoplasms; Leukemia | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Abatacept (Experimental): Participants will receive one of two standard myeloablative conditioning regimens for their stem cell transplant, and will receive an aGvHD prophylaxis regimen including cyclosporine, methotrexate, and abatacept.
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept — Participants will receive one of two standard myeloablative conditioning regimens for their stem cell transplant, and will receive an aGvHD prophylaxis regimen including cyclosporine, methotrexate, and abatacept.
  Other Names: orencia

SUMMARY:
The primary objective of the study is to determine the safety and tolerability when adding abatacept to acute Graft versus Host Disease in transplants for malignant diseases using unrelated donor bone marrow or peripheral blood stem cell grafts.

DETAILED DESCRIPTION:
Acute Graft versus Host Disease (aGvHD) is the most deadly complication facing children who have allogeneic hematopoietic stem cell transplant (HSCT). aGvHD occurs, in large part, because the T cells in the bone marrow graft do not "accept" the presence of the transplant recipient's cells, and mount a severe, debilitating, and often deadly attack against the recipient, striking the skin, the liver, and the gastrointestinal track, most prominently. For patients receiving bone marrow from an unrelated donor, the rate of aGvHD can reach as high as 80%, with up to half of patients dying from this complication. These serious outcomes occur despite our best efforts at aGvHD prevention. Given the lack of success in preventing aGvHD with current therapies, novel therapies to prevent this disease are desperately needed.

In this study, we plan to test a novel drug to prevent aGvHD. This drug, known as abatacept, specifically blocks the activation pathway critical to T cell function known as "T cell costimulation." In particular, it blocks the CD28-mediated costimulation pathway that is critical for optimal T cell activation and proliferation. My research group has done extensive pre-clinical work with this compound. Our work has demonstrated its efficacy in inducing immune tolerance after transplantation in both mouse models and primate models. In addition, patient trials have demonstrated that blocking CD28-directed T cell costimulation can prevent T cell-mediated diseases, including rheumatoid arthritis and psoriasis, and can improve solid organ transplant acceptance. Abatacept is currently FDA approved for use in rheumatoid arthritis. Given this drug's safety and efficacy profile, we have been granted an IND-exemption from the FDA for the inclusion of abatacept in a GvHD-prevention strategy.

This is a safety and tolerability study of the addition of abatacept to a GvHD-prophylaxis regimen. Thus, the primary objective of the study is to determine the safety and tolerability of the addition of abatacept to aGvHD prophylaxis in transplants for malignant hematologic disease using unrelated donor bone marrow or peripheral blood stem cell grafts.

Three secondary objectives will also be addressed:

1. We will estimate the incidence and severity of aGvHD in patients receiving the abatacept-based protocol.
2. We will determine the immune phenotype of donor cells in patients receiving abatacept.
3. We will determine the ability of donor T-cells in patients receiving abatacept to respond to both polyclonal and recipient-specific immune stimulation.

These secondary objectives will allow us to determine the impact of abatacept-containing GvHD prevention on both T cell alloreactivity and on T cell-mediated protective immunity.

This study is for patients older than 12 who have been diagnosed with high-risk leukemia and for whom an unrelated bone marrow transplant is planned. We plan to enroll 10 patients on the study, over a 1-year period from the opening of the trial. Of these ten patients, at least five will be pediatric patients; the other five may be from adult patients taken care of by Winship Cancer Center physicians. All clinical study coordination and biologic studies will be performed by CHOA personnel.

Participants will receive one of two standard myeloablative conditioning regimens for their stem cell transplant, and will receive an aGvHD prophylaxis regimen including cyclosporine, methotrexate, and abatacept. They will have immunologic analysis for 1 year after transplant and clinical analysis for 3 years after transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with AML, with or without a history of myelodysplastic syndrome in one of the following categories.

   (a) Patients in first complete remission with high-risk features
2. Patients with ALL, in either of the following categories:

   1. In 2nd or greater complete remission (complete remission is defined as > 5% blasts in marrow)
   2. Delayed 1st CR-Failure to achieve complete remission after a single round of induction therapy
3. Patients with undifferentiated or biphenotypic leukemia in 1st or greater complete remission.
4. Patients with Myelodysplastic Syndrome(s) with an IPSS score of >1.5 and <10% blasts in the bone marrow at the time of transplant. These conditions will include:

   1. Refractory anemia
   2. Refractory anemia with ringed sideroblasts
   3. Refractory cytopenia with multilineage dysplasia
   4. Refractory cytopenia with multilineage dysplasia and ringed sideroblasts
   5. Refractory anemia with excess blasts-1 (5-10% blasts)
   6. Refractory anemia with excess blasts-2 (10-20% blasts)
   7. Myelodysplastic syndrome, unclassified
   8. MDS associated with isolated del (5q)
   9. Patients diagnosed with AML in CR1 after an initial diagnosis of MDS.
5. Age 12 years or older.
6. No prior allogeneic transplant
7. Karnofsky performance score or Lansky Play-Performance of at least 80.
8. Signed informed consent for adults and for minors the provision of pediatric assent and parental permission.

Exclusion Criteria:

1. Age <12 years old.
2. Patients requiring >2 courses of induction chemotherapy to achieve remission status.
3. HIV infection
4. Tuberculosis Infection
5. Chronic Obstructive Pulmonary Disease
6. Pregnancy (positive serum b-HCG) or breastfeeding
7. Creatinine clearance or nuclear medicine GFR of < 50 mL/min
8. Cardiac ejection fraction < 50%
9. bilirubin > 2 × upper limit of normal or ALT > 4 × upper limit of normal or unresolved veno-occlusive disease.
10. Pulmonary disease with FVC, FEV1 or DLCO parameters <45% predicted (corrected for hemoglobin) or O2 saturation <92% on room air.
11. Karnofsky performance score or Lansky Play-Performance Scale <80
12. Uncontrolled viral, bacterial, or fungal infection at the time of study enrollment
13. Availability of a willing and fully MHC-matched related donor.
14. Positive cytotoxic recipient-donor cross-match or positive HLA antibody screen against donor-disparate antigens.
15. Any active infection.
16. Unable to obtain informed consent.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-11; Primary Completion 2012-11 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Kean, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Koura DT, Horan JT, Langston AA, Qayed M, Mehta A, Khoury HJ, Harvey RD, Suessmuth Y, Couture C, Carr J, Grizzle A, Johnson HR, Cheeseman JA, Conger JA, Robertson J, Stempora L, Johnson BE, Garrett A, Kirk AD, Larsen CP, Waller EK, Kean LS. In vivo T cell costimulation blockade with abatacept for acute graft-versus-host disease prevention: a first-in-disease trial. Biol Blood Marrow Transplant. 2013 Nov;19(11):1638-49. doi: 10.1016/j.bbmt.2013.09.003. Epub 2013 Sep 15. PMID 24047754
- [Result] Suessmuth Y, Mukherjee R, Watkins B, Koura DT, Finstermeier K, Desmarais C, Stempora L, Horan JT, Langston A, Qayed M, Khoury HJ, Grizzle A, Cheeseman JA, Conger JA, Robertson J, Garrett A, Kirk AD, Waller EK, Blazar BR, Mehta AK, Robins HS, Kean LS. CMV reactivation drives posttransplant T-cell reconstitution and results in defects in the underlying TCRbeta repertoire. Blood. 2015 Jun 18;125(25):3835-50. doi: 10.1182/blood-2015-03-631853. Epub 2015 Apr 7. PMID 25852054

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient signed consent but was determined to be an assignment failure prior to starting study activities.
Period: Overall Study
Arm/Group | Abatacept
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Abatacept
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (27)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 8
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Grade III-IV Acute GVHD by Day 100.
Description: Grade III-IV Acute GVHD by Day 100. The incidence of Gr III-IV acute GVHD was measured by the modified Glucksburg scale.
Time Frame: Day 100 post-transplant
Measure: Number; unit: percentage of participants
Arm/Group | Abatacept
Number analyzed (Participants) | 10
percentage of participants | 10

2. Secondary Outcome: Percentage of Participants With Grades III-IV Acute GVHD at 2 Years
Description: The rates of Grades III-IV acute GVHD were measured at 2 years according to standard Glucksberg criteria, which was 10%.
Time Frame: 2 years after transplant
Measure: Number; unit: percentage of participants
Arm/Group | Abatacept
Number analyzed (Participants) | 10
percentage of participants | 10

3. Secondary Outcome: Hematologic and Immunologic Reconstitution
Description: Flow cytometric analysis of CD4 t-cell t-cell reconstitution was performed at day +100 post-transplant.
Time Frame: Day +100 post-transplant
Measure: Mean (Standard Error); unit: cell per microlitre
Arm/Group | Abatacept
Number analyzed (Participants) | 10
cell per microlitre | 285 (105)

4. Secondary Outcome: Protective Immunity
Description: Percent of CMV virus binding CD8+ t-cells at day +365 post-transplant
Time Frame: Day +365 post-transplant
Measure: Mean (Standard Error); unit: percentage of total CD8+ t-cells
Arm/Group | Abatacept
Number analyzed (Participants) | 10
percentage of total CD8+ t-cells | 2.8 (1.7)

ADVERSE EVENTS:
Time Frame: One year post-transplant.
Description: Attribution of adverse events when patients are co-enrolled on other trials: because abatacept's effects are strictly immunologic and because co-enrollment will only be allowed in trials testing agents without immunomodulatory effects, all adverse events stemming directly or indirectly from immune deficiency or immune dysregulation will be attributed (definite, probable or possible depending on the circumstances) to abatacept and not the agent being tested in the other trial.
Groups:
- Abatacept: In this trial, we will test the safety and tolerability of the addition of the CD28-B7 blockade agent, abatacept, as an adjunctive therapy for the prevention of GvHD in a high-risk BMT cohort. Four doses of abatacept will be given according to a dosing schedule based on previous trials using CD28-B7 blockade with belatacept in kidney transplantation. Pharmacokinetic and pharmakodynamic analysis of abatacept will be undertaken, as well as an evaluation of the incidence and severity of acute GvHD in this patient cohort.
  Dosage: Abatacept is administered as an intravenous infusion under medically controlled conditions. Dose is 10mg/kg with a maximum dose of 1 gram. Abatacept should be administered as a 30-minute intravenous infusion. In this study, abatacept will be dosed on days -1, +5, +14, +28 post-transplant. Small adjustments in dose to accommodate abatacept vial size may be acceptable. These dose adjustments must be approved by the study PI.
Arm/Group | Abatacept
Serious Adverse Events (participants affected / at risk) | 7/10
Other Adverse Events (participants affected / at risk) | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abatacept (N=10)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4)
Bacteremia with coagulase negative staphylococcus (Infections and infestations) | 1 (2)
Upper Respiratory Infection - Parainfluenza (Infections and infestations) | 1 (1)
Bacteremia with E. coli (Infections and infestations) | 1 (1) — i
Upper Respiratory Infection - Rhinovirus (Infections and infestations) | 1 (1)
Perianal cellulitis (Infections and infestations) | 1 (1)
Hemorrhagic cystitis with BK virus (Infections and infestations) | 1 (1)
Polyclonal lymphoproliferative disorder (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abatacept (N=10)
Renal toxicity (Renal and urinary disorders) | 4 (4) — Renal toxicity grade 2
Mucositis oral (Gastrointestinal disorders) | 5 (5) — Mucositis oral grade 2
Bladder toxicity (Infections and infestations) | 1 (1) — bladder grade 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No